CLINICAL TRIAL: NCT03588338
Title: The Effect of Paracetamol on Postoperative Nausea and Vomiting Following Maxillofacial Surgery: a Prospective, Randomised, Double-blind Study
Brief Title: Paracetamol on Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Ozlem Kocaturk, Faculty of Dentisty Oral and Maxillofacial Surgery, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017/1081
Record Dates: First submitted 2018-07-05; First posted 2018-07-17 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: PONV; Paracetamol
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Acetaminophen; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perfalgan (Active Comparator): 1.5 mg/kg intravenous, intraoperative (20 min before end of the surgery)
  Interventions: Drug: Perfalgan; Drug: Control
- Control (Other): 1.5 mg/kg intravenous, intraoperative (20 min before end of the surgery)
  Interventions: Drug: Perfalgan; Drug: Control

INTERVENTIONS:
Drug: Perfalgan — For postoperative pain
  Other Names: Paracetamol
Drug: Control — For postoperative nausea and vomiting
  Other Names: Saline

SUMMARY:
The drugs with both high potency and low side effects are preferred in the prevention of postoperative nausea and vomiting (PONV) which is a common problem. This prospective randomized study aimed to compare the efficacy of paracetamol on PONV in adults undergoing maxillofacial surgery.

DETAILED DESCRIPTION:
One hundred-twenty patients are randomly divided into two groups; the paracetamol group who received the IV infusion of paracetamol (1.5 ml/kg); and the metoclopramide group who received the IV infusion of saline (1.5 mg/kg). The presence of vomiting and the actions indicative of nausea, such as repeated gagging or spitting, within 24h following general anesthesia are defined as PONV. All PONV episodes and postoperative pain scores are recorded during 24h postoperatively. The postoperative 0-4h and 4-24h are defined as early and late postoperative period, respectively. Intravenous 4 mg ondansetron as rescue antiemetic drug is administered in case of two or more vomiting episodes.

ELIGIBILITY:
Inclusion Criteria:

* ASA (the classification of the American Society of Anesthesiologists) physical status I-II
* Patients who scheduled for elective maxillofacial surgery under general anesthesia

Exclusion Criteria:

* Patients with a history of allergy to any of the study medications (opioid, general anesthetic agents or paracetamol)
* History of opioid use, hepatic or renal disease, coronary, psychotic and neurologic diseases
* Use of antiemetic, antihistaminic, analgesic or corticosteroid 24 hours (h) prior to surgery

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Preventing of postoperative nausea and vomiting | First 24 hours postoperatively
  Preventing of postoperative nausea and vomiting in postoperative care unit

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Menderes University, Study Director — Aydin Adnan Menderes University
Locations (1):
- Ozlem Kocaturk, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cok OY, Eker HE, Pelit A, Canturk S, Akin S, Aribogan A, Arslan G. The effect of paracetamol on postoperative nausea and vomiting during the first 24 h after strabismus surgery: a prospective, randomised, double-blind study. Eur J Anaesthesiol. 2011 Dec;28(12):836-41. doi: 10.1097/EJA.0b013e32834c580b. PMID 21986980